CLINICAL TRIAL: NCT07320820
Title: Assessment of Quality of Life, Patient Satisfaction, Swallowing Function, Voice Outcomes, Pain, and Anxiety-Depression at Baseline and at 3-, 6-, and 12-Month Follow-Up in Patients Diagnosed With Laryngeal Squamous Cell Carcinoma: A Prospective Questionnaire-Based Study
Brief Title: Quality of Life and Functional Outcomes in Laryngeal Cancer Patients
Acronym: QoL in LSSC
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sumeyra DOLUOGLU, Associate Professor, Saglik Bilimleri Universitesi
Other Study IDs: SaglikBUniversity; Ankara Etlik City Hospital (Registry Identifier: Sumeyra Doluoglu)
Record Dates: First submitted 2025-12-13; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Laryngeal Carcinoma; Quality of Life (QOL); Patient Satisfaction; Voice Quality; Swallowing Function; Pain Management; Anxiety Depression
MeSH Terms: conditions — Laryngeal Neoplasms; Patient Satisfaction; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Surgical Treatment Group: This group includes patients with laryngeal squamous cell carcinoma who undergo primary surgical treatment, such as partial or total laryngectomy, with or without neck dissection, in accordance with standard oncological indications. Patients in this group may receive adjuvant radiotherapy or chemoradiotherapy when clinically indicated based on pathological findings.
  Interventions: Other: Quality of Life Assessment; Other: Patient Satisfaction Assessment; Other: Swallowing Function Assessment; Other: Voice Assessment; Other: Pain Assessment; Other: Anxiety and Depression Assessment
- Radiotherapy Group: This group consists of patients with laryngeal squamous cell carcinoma treated with definitive radiotherapy as the primary treatment modality. Radiotherapy is delivered according to established clinical protocols, and no surgical intervention to the primary tumor is performed as the initial treatment.
  Interventions: Other: Quality of Life Assessment; Other: Patient Satisfaction Assessment; Other: Swallowing Function Assessment; Other: Voice Assessment; Other: Pain Assessment; Other: Anxiety and Depression Assessment
- Chemoradiotherapy Group: This group includes patients with laryngeal squamous cell carcinoma who receive concurrent chemoradiotherapy as the primary treatment modality, typically for organ preservation purposes or in locally advanced disease. Chemotherapy is administered concurrently with radiotherapy in accordance with institutional and international treatment guidelines.
  Interventions: Other: Quality of Life Assessment; Other: Patient Satisfaction Assessment; Other: Swallowing Function Assessment; Other: Voice Assessment; Other: Pain Assessment; Other: Anxiety and Depression Assessment

INTERVENTIONS:
Other: Quality of Life Assessment — Quality of life will be assessed using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) and the Head and Neck Cancer-Specific Module (QLQ-H&N35). The QLQ-C30 evaluates global health status, functional domains, and symptom scales, while the QLQ-H&N35 provides disease-specific information related to head and neck cancer, including symptoms associated with swallowing, speech, pain, and social eating.
Other: Patient Satisfaction Assessment — Patient satisfaction with cancer care will be evaluated using the EORTC In-Patient Satisfaction with Care Questionnaire (PATSAT-C33). This instrument assesses patients' perceptions of the quality of care, communication with healthcare professionals, and overall satisfaction with treatment and supportive care services.
Other: Swallowing Function Assessment — Swallowing function will be assessed using the MD Anderson Dysphagia Inventory (MDADI) and the Eating Assessment Tool-10 (EAT-10). The MDADI is a disease-specific, patient-reported outcome measure that evaluates the impact of dysphagia on quality of life across emotional, functional, and physical domains. The EAT-10 is a symptom-specific screening tool designed to quantify the severity of swallowing difficulties and their effect on daily activities.
Other: Voice Assessment — Voice-related outcomes will be evaluated using the Voice Handicap Index-10 (VHI-10), a validated patient-reported questionnaire that measures the perceived impact of voice disorders on functional, physical, and emotional aspects of daily life.
Other: Pain Assessment — Pain intensity will be assessed using the Visual Analog Scale (VAS), a widely used, validated tool that allows patients to rate their pain severity on a continuous scale, providing a quantitative measure of pain perception over time.
Other: Anxiety and Depression Assessment — Psychological status will be evaluated using the Hospital Anxiety and Depression Scale (HADS), a validated self-report instrument designed to assess symptoms of anxiety and depression in medically ill populations, minimizing the influence of somatic symptoms related to physical illness.

SUMMARY:
Laryngeal squamous cell carcinomas are head and neck malignancies that directly affect both swallowing and voice functions and are associated with a significant deterioration in patients' quality of life throughout the treatment process.

The aim of this study is to evaluate quality of life, voice and swallowing functions, pain, anxiety-depression levels, and patient satisfaction at the pre-treatment period and at the 3rd, 6th, and 12th months post-treatment in patients with laryngeal malignancies, using validated questionnaires, in order to:

Elucidate the course of functional recovery following treatment,

Individualize rehabilitation and follow-up strategies, and

Examine the relationship between functional outcomes and oncological survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of enrollment.
* Histopathologically confirmed diagnosis of laryngeal squamous cell carcinoma.
* Planned to undergo surgical treatment or radiotherapy/chemoradiotherapy as part of standard oncological care.
* Willing and able to participate in the study and to provide written informed consent.
* No history of psychiatric or neurological disorders that could impair comprehension, questionnaire completion, or study participation.

Exclusion Criteria:

* Age < 18 years.
* Presence of comorbid conditions that may independently affect swallowing or voice functions.
* Patients who withdraw consent or request to discontinue participation during or after the treatment period.
* History of psychiatric disorders or use of psychiatric medications that may interfere with study participation or completion of patient-reported outcome measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with laryngeal squamous cell carcinoma who are planned to undergo surgical treatment, radiotherapy, or chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Head and Neck-Specific Quality of Life (EORTC QLQ-H&N35) | Baseline (pre-treatment), 3 months, 6 months, and 12 months after completion of treatment. Type of Measure: Patient-reported outcome; continuous scale.
  Change in head and neck cancer-specific quality of life as assessed by the EORTC QLQ-H&N35 questionnaire. The instrument evaluates symptoms and functional impairments related to head and neck cancer and its treatment; higher scores indicate greater symptom burden and worse quality of life.

SECONDARY OUTCOMES:
Change in Global Quality of Life (EORTC QLQ-C30) | Baseline, 3 months, 6 months, and 12 months after completion of treatment.
  Change in global health status/quality of life score measured by the EORTC QLQ-C30 questionnaire. Higher scores on the global health status scale indicate better overall quality of life.
Change in Swallowing Function (MD Anderson Dysphagia Inventory - MDADI) | Baseline, 3 months, 6 months, and 12 months after completion of treatment.
  Change in swallowing-related quality of life assessed by the MD Anderson Dysphagia Inventory (MDADI). Higher scores indicate better perceived swallowing function and quality of life.
Change in Patient Satisfaction (EORTC PATSAT-C33) | 3 months, 6 months, and 12 months after completion of treatment.
  Change in patient satisfaction with cancer care measured using the EORTC PATSAT-C33 questionnaire, which assesses satisfaction with physicians, nurses, organization of care, and overall treatment experience. Higher scores indicate greater patient satisfaction.
Change in Dysphagia Severity (Eating Assessment Tool - EAT-10) | Baseline, 3 months, 6 months, and 12 months after completion of treatment.
  Change in dysphagia symptom severity measured by the Eating Assessment Tool-10 (EAT-10). Higher scores indicate more severe swallowing difficulties.
Change in Voice-Related Handicap (Voice Handicap Index-10 - VHI-10) | Baseline, 3 months, 6 months, and 12 months after completion of treatment.
  Change in patient-perceived voice handicap measured by the Voice Handicap Index-10 (VHI-10). Higher scores indicate greater perceived voice-related disability.
Change in Pain Intensity (Visual Analog Scale - VAS) | Baseline, 3 months, 6 months, and 12 months after completion of treatment.
  Change in pain intensity measured using a Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity.
Change in Anxiety and Depression Levels (Hospital Anxiety and Depression Scale - HADS) | Baseline, 3 months, 6 months, and 12 months after completion of treatment.
  Change in anxiety and depression symptoms measured by the Hospital Anxiety and Depression Scale (HADS), including HADS-Anxiety (HADS-A) and HADS-Depression (HADS-D) subscales. Higher scores indicate greater psychological distress.

IPD SHARING:
Plan to Share IPD: No